CLINICAL TRIAL: NCT07318259
Title: Study of Ultra-Fast Autologous BCMA/CD70-Targeted Chimeric Antigen Receptor T (CAR- T) Therapy for Refractory Systemic Lupus Erythematosus
Brief Title: Study of Ultra-Fast BCMA/CD70 CAR-T Therapy for Refractory SLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC093
Record Dates: First submitted 2025-12-11; First posted 2026-01-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: BCMA/CD70; CAR-T
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: Treatment of patients with refractory systemic lupus erythematosus using ultra-fast BCMA/CD70-targeted CAR-T cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): This trial was designed as an open, single-arm, single-center, dose-increasing trial.
  Interventions: Biological: BCMA/CD70 CAR-T cells

INTERVENTIONS:
Biological: BCMA/CD70 CAR-T cells — Three dose groups (1.5×10^5/kg, 5×10^5/kg, 10×10^5/kg) were set up, starting from the low dose group climbing to explore the safe and effective dose.

SUMMARY:
This is an investigator-initiated trial aimed at assessing the safety and efficacy of ultra-fast autologous BCMA/CD70-targeted CAR-T cells in the treatment of refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a serious autoimmune disease that can lead to extensive damage in multiple organs and systems, ultimately resulting in disability and even death.

Currently, the primary treatment for SLE relies on glucocorticoids and immunosuppressants to alleviate symptoms. However, due to the absence of a curative treatment, patients typically need to remain on medication indefinitely. In recent years, biological agents such as belimumab and rituximab have been introduced for the treatment of SLE, but these treatments cannot completely eliminate autoimmune B cells in the bone marrow, leading to unsatisfactory overall outcomes. Furthermore, discontinuing these drugs can lead to disease relapse, and there is still no cure for SLE, leaving patients facing the challenges of lifelong medication and an incurable disease.

CAR-T therapy is an adoptive cell therapy that uses genetic modification technology to reprogram T cells and eliminate target cells expressing disease-related antigens through antigen-specific recognition. Since 2019, CAR-T cell therapy has been successfully applied to autoimmune diseases. Clinical studies have demonstrated that CAR-T cells hold significant therapeutic potential for SLE. Compared with traditional CAR-T cells, ultra-fast CAR-T, relying on an innovative CAR-T manufacturing system, can produce CAR-T cells in an extremely short period of time (with a preparation time of only 10 minutes).

The purpose of this study is to assess the safety and efficacy of the ultra-fast autologous BCMA/CD70-targeted CAR-T cells in the treatment of refractory SLE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Diagnosed with SLE according to the 2019 EULAR/ACR SLE classification criteria, and still in moderate to severe disease activity despite ≥3M of high dose glucocorticoids(prednisone≥1mg/kg/d or other equivalent amount of other steriod), and/or hydroxychloroquine, and at least 2 DMARDs(include cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, cyclosporin, tacrolimus, sirolimus, leflunomide, telitacicept, beliumab, and rituximab) or intolerant to standard treatments;
* SLEDAI-2K score ≥ 8 points;
* Meet the standards of leukapheresis or intravenous blood collection, and no contraindication for leukapheresis;
* Negative pregnancy test for female subjects of childbearing age, and agree to take effective contraceptive measures until one year after CAR-T infusion;
* Participant or his/her guardians agree to participate in the clinical trial and sign the informed consent form which indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

* Central nervous system (CNS) disease: CNS neurolupus requires intervention within 30 days;
* Have a history of congenital heart disease or acute myocardial infarction within 6 months prior to screening or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia, etc.); or NYHA classification class IV; or combined with moderate to massive pericardial effusion, serious myocarditis, etc; or patient with unstable vital signs who need hypertensive drugs;
* The functions of important organs meet one of the following conditions: (1)renal function: eGFR<30mL/min/1.73m2 or require renal replacement therapy; (2)liver function: AST and ALT>3.0 ULN, total Bilirubin (TBIL) in serum >2.0×ULN; (3)lung function: SpO2<92% with no oxygen inhalation;
* Uncontrollable infection or active infection that requires systemic treatment within 3 months prior to screening;
* Received hematopoietic stem cell transplantation within 3 months prior to screening, or ≥Grade 2 GVHD within 2 weeks prior to screening;
* Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; or positive for human immunodeficiency virus (HIV) antibodies; or syphilis test positive;
* Suffered from active pulmonary tuberculosis at screening;
* Received live vaccine within 4 weeks prior to screening;
* Positive in blood pregnancy test;
* Suffered from malignant disease such as tumors (excluding tumors without active lesions and ending treatment for more than 5 years, as well as fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, thyroid cancer after radical resection, ductal carcinoma in situ after radical resection);
* Patients who participated in other clinical study within 3 months prior to screening;
* Any other conditions that the investigators deem it unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
The safety of CAR-T cell therapy in patients with refractory SLE [Safety] | 3 months
  Types, frequency and severity of adverse events.
The changes from baseline in SLEDAI-2K [efficacy] | 6 months
  Systemic Lupus Erythematosus Disease Activity Index 2000(SLEDAI-2K) is from 0 to 105 points. The higher score means the stronger disease activity.
The changes from baseline in PGA [efficacy] | 6 months
  Physician Global Assessment(PGA) is a continuous visual analogue scale with 0, 1, 2, and 3 scales. "0" indicates no disease activity and "3" indicates the most severe disease activity.
The changes from baseline in BILAG-2004 [efficacy] | 6 months
  British Isles Lupus Assessment Group Index 2004(BILAG-2004) consists of 8 systems, each of which is classified as A, B, C and D respectively. "A" indicates that the condition is highly active and requires active treatment. "B" indicates that the condition is active and requires close monitoring or symptomatic treatment. "C" indicates a stable condition. "D" indicates that the system is not involved.
The number of patients with SRI-4 response [efficacy] | 3 months
  The definition of SRI-4 response: SLEDAI-2K ≥ 4-Point improvement; PGA with no worsening (<0.3 point increase); BILAG 2004 with no new A domain score and no more than 1 new B domain scores.
The number of patients with LLDAS [efficacy] | 6 months
  The definition of LLDAS: SLEDAI-2K ≤ 4 and no disease activity in major organs (kidneys, central nervous system, heart and lungs), and no vasculitis or fever; no new disease activity symptoms were added compared with previous disease assessments; PGA ≤ 1; irrespective of serology; with permitted use of low-dose glucocorticoids (prednisolone ≤ 7.5 mg/day), and/or stable immunosuppressives and biologics.
The number of patients with DORIS [efficacy] | 6 months
  The definition of DORIS: SLEDAI-2K = 0 ; PGA < 0.5 ; irrespective of serology; with permitted use of antimalarials, low-dose glucocorticoids (prednisolone ≤ 5 mg/day), and/or stable immunosuppressives and biologics.

SECONDARY OUTCOMES:
The changes of anti-ds-DNA antibody after infusion [efficacy] | 6 months
The changes of 24h urine protein after infusion [efficacy] | 6 months
The changes of serum complement C3 and C4 after infusion [efficacy] | 6 months
Cmax of CAR-T cells [PK parameter] | 3 months
  The peak plasma concentration (Cmax) of amplified CAR-T cells in peripheral blood after infusion.
Tmax of CAR-T cells [PK parameter] | 3 months
  The time of amplified CAR-T cells in peripheral blood to reach the maximum concentration (Tmax).
AUC28d/90d of CAR-T cells [PK parameter] | 3 months
  The area under the plasma concentration-time curve from 28 to 90 days after infusion (AUC28d/90d).
The degree of B cell and T cell depletion [PD parameter] | 3 months
  The degree of B cell and T cell depletion at various time points.
The concentration levels of IL-6 [PD parameter] | 3 months
  CAR-T-related serum cytokines such as IL-6.
The concentration levels of CRP [PD parameter] | 3 months
The concentration levels of ferritin [PD parameter] | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China